CLINICAL TRIAL: NCT00158626
Title: A Feasibility Study for an RCT of a Pelvic Floor Muscle Training Intervention for Pelvic Organ Prolapse
Brief Title: Does Doing Pelvic Floor Exercise Ease Symptoms for Women Living With Prolapse?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZH/4/95; NRR N0470119684;; ISRCTN44995705
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Uterine Prolapse
Keywords: physical therapy; physiotherapy; pelvic organ prolapse
MeSH Terms: conditions — Uterine Prolapse; Pelvic Organ Prolapse

INTERVENTIONS:
Behavioral: pelvic floor muscle training

SUMMARY:
The purpose of this study is to investigate the feasibility of undertaking a multi-centre randomised controlled trial of the effectiveness of a pelvic floor muscle training (PFMT) intervention for women with pelvic organ prolapse.

DETAILED DESCRIPTION:
Pelvic organ prolapse is a common female condition; it is estimated that 50% of women experience some degree of prolapse and 30% of attendees at gynaecology clinics present with this problem. Vaginal delivery is cited as the main cause of prolapse but menopause, heavy lifting, chronic cough and straining are also important factors. Symptoms associated with prolapse are backache, pelvic heaviness and bladder, bowel and sexual dysfunction. Thus, the condition is debilitating and can greatly affect the sufferer's daily activities and quality of life.

Traditionally, treatment of prolapse consists of surgery or conservative treatment. Surgical procedures to repair the fascia vary and improved techniques are constantly being sought. At present however the recurrence rate of prolapse after surgery is 25%, with 80% re-occurring within two years of surgery. Conservative treatment is often considered if the prolapse is small or the patient is not a good candidate for surgery. There are three types of conservative treatment: 1) Physical interventions that aim to improve pelvic floor muscle function by using pelvic floor muscle assessment and exercises, neuromuscular electrical stimulation, 2) Mechanical interventions that aim to manage the prolapse by supporting the pelvic area (e.g. using vaginal ring pessaries) and, 3) Lifestyle interventions (such as weight loss and reducing exacerbating activities) that seek to avoid exacerbation of the prolapse by decreasing intra-abdominal pressure.

The promotion of pelvic floor exercises (PFEs) for prolapse varies between hospitals with some providing only a patient information leaflet and others giving individual instruction from a physiotherapist. Such a programme is referred to as pelvic floor muscle training (PFMT). An ongoing Cochrane review of the literature has, to date, found no evidence for management of pelvic organ prolapse using PFMT. This proposal addresses a gap in the research evidence by developing a multi-centre randomised controlled trial of a PFMT intervention for women with prolapse. The feasibility of all aspects of such a trial will be assessed, and pilot data will be collected at two Scottish Centres (Glasgow and Aberdeen). Ultimately, a multi-centre trial would aim to establish if PFMT is better than standardised management for reducing prolapse specific symptoms, prolapse severity, the need for surgical prolapse repair and the costs associated with the condition.

50 women attending out-patient clinics who are suitable for the study will be randomised to either the control or intervention arm of the trial. Women in the intervention arm will receive an individualised programme of PFMT delivered by a physiotherapist via 5 sessions of physiotherapy over a 16 week period. This programme will include pelvic muscle assessment, teaching and prescription of pelvic floor exercises, and provision of lifestyle advice. Women in the control arm will only receive, by post, a lifestyle advice leaflet. Type and severity of prolapse will be quantified according to ICS guidelines (POP-Q method). Data on outcome measures relating to improvement in prolapse symptoms and associated quality of life will be obtained via self-completion questionnaires

ELIGIBILITY:
Inclusion Criteria:

* women with previously untreated stage I or II pelvic organ prolapse attending gynaecology, urogynaecology and prolapse specific out-patient clinics at South Glasgow University NHS Trust and Grampian University Hospitals NHS Trust

Exclusion Criteria:

* previous surgical or conservative treatment for prolapse (e.g. pessary management or previous pelvic floor muscle training)
* women considered not suitable for physiotherapy treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change in prolapse related symptoms and associated quality of life measured by a combination of ICIQ tools, the Prolapse Quality of Life tool and study specific questions at baseline, 20 weeks and 26 weeks.

SECONDARY OUTCOMES:
Change in prolapse severity using the POP-Q method of quantification at baseline and 20 weeks, days of symptoms at baseline and 26 weeks, and general health status (SF-12) at baseline, 20 weeks and 26 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Hagen, Principal Investigator — NMAHP Reserach Unit, Glasgow Caledonian University
Locations (2):
- United Kingdom (2):
  - Grampian University Hospitals, NHS Grampian, Aberdeen
  - South Glasgow University Hospitals Division, NHS Greater Glasgow, Glasgow

REFERENCES:
- [Background] Hagen S, Stark D, Glazener C, Sinclair L, Ramsay I. A randomized controlled trial of pelvic floor muscle training for stages I and II pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):45-51. doi: 10.1007/s00192-008-0726-4. Epub 2008 Sep 20. PMID 18806910
- See also: results paper in IUJ — http://link.springer.com/article/10.1007/s00192-008-0726-4#